CLINICAL TRIAL: NCT00317681
Title: The Efficacy of Topical Tacrolimus in the Treatment of Cutaneous Lupus Erythematosus - a Multi-Center-Trial
Brief Title: Efficacy of Topical Tacrolimus in Different Subtypes With Cutaneous Lupus Erythematosus (CLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AMG 001; 2004-005020-41
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: Cutaneous lupus erythematosus; Tacrolimus ointment; Topical treatment; Skin lesions
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

INTERVENTIONS:
Drug: Tacrolimus ointment

SUMMARY:
The purpose of this study is to evaluate the efficacy of topical tacrolimus in different subtypes of cutaneous lupus erythematosus. As shown by several groups activated memory T lymphocytes play a key role in the pathogenesis of lupus erythematosus. Tacrolimus targets T lymphocytes and suppresses their activation by inhibiting the expression of cytokine genes, such as IL-2. Therefore, treatment of cutaneous lupus erythematosus with topical tacrolimus might result in an improvement of skin lesions in such patients.

DETAILED DESCRIPTION:
In patients with cutaneous lupus erythematosus (CLE), topical corticosteroids are the mainstay of treatment; however, a long-term use can lead to numerous side effects including skin atrophy. Recently, topical tacrolimus has been suggested to be effective in patients with different manifestations of CLE as single or additive therapy. Its anti-inflammatory effect can be explained by inhibition of calcineurin and suppression of proinflammatory cytokines such as interleukins-2, -3, -4, granulocyte colony-stimulating factor, and tumour necrosis factor alpha. In this study, we evaluate the efficacy of tacrolimus in 30 patients with different forms of CLE (ACLE, SCLE, DLE, LET). During a period of 3 months tacrolimus ointment and its placebo are applied on two separate skin lesions. Clinical follow-up examinations including photo documentation are performed every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous lupus erythematosus confirmed by histological analysis
* Topical use of glucocorticosteroids stopped at least two weeks before the start of the study
* Presence of two primary skin lesions with a clinical score ≥ 1
* Written informed consent available prior to any screening procedures

Exclusion Criteria:

* Systemic medication if taken for lupus erythematosus (e.g. chloroquine or hydroxychloroquine) started at least 6 months prior to the beginning of the study
* Women of childbearing potential using inadequate birth control measures
* Pregnancy and lactation
* Known hypersensitivity to tacrolimus or any of the excipients
* Patients receiving systemic immunosuppressive drugs and cytotoxic agents other than antimalarial agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-08; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Difference in skin lesions of patients with CLE before (begin of study) and after treatment (end of study) evaluated by a clinical score

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, MD, Principal Investigator — Heinrich-Heine-University of Duesseldorf, Department of Dermatolgy
Locations (1):
- Heinrich-Heine-University of Duesseldorf, Department of Dermatology, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Bacman D, Tanbajewa A, Megahed M, Ruzicka T, Kuhn A. [Topical treatment with tacrolimus in lupus erythematosus tumidus]. Hautarzt. 2003 Oct;54(10):977-9. doi: 10.1007/s00105-003-0593-3. No abstract available. German. PMID 14513247
- [Background] Kuhn A, Gensch K, Stander S, Bonsmann G. [Cutaneous lupus erythematosus. Part 2: diagnostics and therapy]. Hautarzt. 2006 Apr;57(4):345-8; quiz 359. doi: 10.1007/s00105-006-1138-3. German. PMID 16547761
- [Background] Kuhn A, Gensch K, Stander S, Bonsmann G. [Cutaneous lupus erythematosus. Part 1: clinical manifestations and classification]. Hautarzt. 2006 Mar;57(3):251-67; quiz 268. doi: 10.1007/s00105-006-1094-y. German. PMID 16501922